CLINICAL TRIAL: NCT03709225
Title: Exploring the Feasibility of a Mindfulness-Music Intervention to Reduce Anxiety and Stress in Adolescents and Young Adults Receiving Cancer Treatment
Brief Title: Mindfulness-Music Intervention for Adolescents and Young Adults With Cancer
Acronym: MAYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Robert Knoerl, PhD, RN, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-341
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Anxiety; Oncology; Stress
Keywords: Anxiety; Music Therapy; Oncology; Adolescent and Young Adults
MeSH Terms: conditions — Anxiety Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music-based meditation (Experimental): The music therapy intervention consists of four in-person sessions (45 minutes) over twelve weeks. Content includes:
  * Introduction to music therapy and mindfulness
  * Music-based meditation
  * Using personal music to shift energy, mood, and support relaxation
  * Mindfulness through active music making
  * Discuss bringing mindfulness to daily activities
  Interventions: Behavioral: Music-based meditation

INTERVENTIONS:
Behavioral: Music-based meditation — The program is designed to incorporate music-based meditation practices and music making activities (e.g., guitar, drums) to help promote relaxation during cancer treatment

SUMMARY:
This study is evaluating how well a music therapy program works to improve anxiety and stress in adolescents and young adults receiving cancer treatment.

DETAILED DESCRIPTION:
This research study will test how well a music therapy program works to improve anxiety and stress in adolescents and young adults receiving cancer treatment. The program is designed to incorporate music-based meditation practices and music making activities (e.g., guitar, drums) to help promote relaxation during cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 - 39 years of age
* Have a diagnosis of any cancer
* Have begun treatment for cancer and plan to receive active cancer treatment (e.g., radiation, chemotherapy, or oral chemotherapy) over the next eight weeks
* Signed informed consent/assent
* Willingness to participate in all study activities
* Speak/read English

Exclusion Criteria:

* Prognosis < 3 months,
* Self-report inability to physically interact with musical instruments (e.g., hold instruments)
* Documentation of significant hearing impairment (e.g., deaf).

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Number of adolescent and young adults recruited to participate in the music therapy program | From enrollment to end of treatment at 12 weeks
  Feasibility of participant recruitment to the music intervention
Frequency of music therapy sessions attended by participants | From enrollment to end of treatment at 12 weeks
  Feasibility of participant adherence to the music intervention
Frequency of outcome assessments completed by participants. | From enrollment to end of treatment at 12 weeks
  Feasibility of participant adherence to outcome assessments

SECONDARY OUTCOMES:
Acceptability and Satisfaction with Participation in Music Therapy Intervention as measured by the Adapted Acceptability E - Scale. | End of treatment at 12 weeks
  Each item of the Adapted Acceptability E - Scale is scored individually on a 1 - 5 scale, with higher scores representing greater acceptability and satisfaction with the music therapy intervention.
Post-traumatic growth | From enrollment to end of treatment at 12 weeks
  Change in Post Traumatic Growth Inventory - Short Form score from enrollment to the end of treatment at 12 weeks. Total scores on the Post Traumatic Growth Inventory Short Form range from 0 - 50, with higher scores representing greater post-traumatic growth.
Stress | From enrollment to end of treatment at 12 weeks
  Change in Perceived Stress Scale score from enrollment to the end of treatment at 12 weeks. The scale is scored from 0 - 40, with higher scores representing greater stress.
Pain Interference: PROMIS | From enrollment to end of treatment at 12 weeks
  Change in Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference 4a score from enrollment to the end of treatment at 12 weeks. Total scores range from 41.6 - 75.6, with higher scores representing worse pain interference.
Fatigue | From enrollment to end of treatment at 12 weeks
  Change in Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue 4a score from enrollment to the end of treatment at 12 weeks. Total scores range from 33.7 - 75.8, with higher scores representing worse fatigue.
Satisfaction with participation in social roles: PROMIS | From enrollment to end of treatment at 12 weeks
  Change in Patient Reported Outcomes Measurement Information System (PROMIS) Satisfaction with Participation in Social Roles 4a score from enrollment to end of treatment at 12 weeks. Total scores range from 29 - 64.1, with higher scores representing worse satisfaction with participation in social roles.
Pain Intensity: PROMIS | From enrollment to end of treatment at 12 weeks
  Change in 0 - 10 numerical rating scale of average pain (included in Patient Reported Outcomes Measurement Information System (PROMIS) - 29 profile)) from enrollment to end of treatment at 12 weeks. Total scores range from 0 - 10, with higher scores representing worse pain.
Depression | From enrollment to end of treatment at 12 weeks
  Change in Patient Reported Outcomes Measurement Information System (PROMIS) Depression 4a score from enrollment to the end of treatment at 12 weeks. Total scores range from 41.0 - 79.4, with higher scores representing worse depression.
Anxiety | From enrollment to end of treatment at 12 weeks
  Change in Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety 4a score from enrollment to the end of treatment at 12 weeks. Total scores range from 40.3 - 81.6, with higher scores representing worse anxiety.
Physical Function | From enrollment to end of treatment at 12 weeks
  Change in Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function 4a score from enrollment to the end of treatment at 12 weeks. Total scores range from 22.9 - 56.9, with higher scores representing worse physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knoerl, PhD, RN, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knoerl R, Mazzola E, Woods H, Buchbinder E, Frazier L, LaCasce A, Luskin MR, Phillips CS, Thornton K, Berry DL, Ligibel J. Exploring Influencing Factors of Anxiety Improvement Following Mindfulness-Based Music Therapy in Young Adults with Cancer. J Music Ther. 2023 Jun 3;60(2):131-148. doi: 10.1093/jmt/thac017. PMID 36787235
- [Derived] Phillips CS, Bockhoff J, Berry DL, Buchbinder E, Frazier AL, LaCasce A, Ligibel J, Luskin MR, Woods H, Knoerl R. Exploring Young Adults' Perspectives of Participation in a Mindfulness-Based Music Therapy Intervention Before and During the COVID-19 Pandemic. J Adolesc Young Adult Oncol. 2023 Aug;12(4):569-576. doi: 10.1089/jayao.2022.0090. Epub 2023 Feb 8. PMID 36752714
- [Derived] Knoerl R, Mazzola E, Woods H, Buchbinder E, Frazier L, LaCasce A, Li BT, Luskin MR, Phillips CS, Thornton K, Berry DL, Ligibel JA. Exploring the Feasibility of a Mindfulness-Music Therapy Intervention to Improve Anxiety and Stress in Adolescents and Young Adults with Cancer. J Pain Symptom Manage. 2022 Apr;63(4):e357-e363. doi: 10.1016/j.jpainsymman.2021.11.013. Epub 2021 Dec 8. PMID 34896280
- [Derived] Knoerl R, Phillips CS, Berfield J, Woods H, Acosta M, Tanasijevic A, Ligibel J. Lessons learned from the delivery of virtual integrative oncology interventions in clinical practice and research during the COVID-19 pandemic. Support Care Cancer. 2021 Aug;29(8):4191-4194. doi: 10.1007/s00520-021-06174-0. Epub 2021 Mar 26. PMID 33772364

DOCUMENTS (1):
  • Informed Consent Form (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT03709225/ICF_000.pdf